CLINICAL TRIAL: NCT04282967
Title: IIT2019-14-SHIRAZIP-SWEAT: Streaming Web-based Exercise At Home: A Pilot Study
Brief Title: Streaming Web-based Exercise At Home: A Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Celina Shirazipour (Other)
Responsible Party: Sponsor-Investigator, Celina Shirazipour, Assistant Professor, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2019-14-SHIRAZIP-SWEAT
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer; Breast Cancer Female
Keywords: Exercise; Breast Cancer Survivor; Prostate Cancer Survivor
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): For the first 12 weeks on study (Part 1), participants will train with an exercise physiologist (EP) for 150 minutes/week. This training will be delivered by web-based video conferencing. For the next 12 weeks (Part 2), participants will be instructed to do patient-directed exercise.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — For the first 12 weeks on study (Part 1), participants will train with an exercise physiologist for 150 minutes/week. This training will be delivered by web-based video conferencing. For the next 12 weeks (Part 2), participants will be instructed to do patient-directed exercise.

SUMMARY:
This is a single-arm pilot study to evaluate the use of web-based video conferencing as a method of exercise training delivery. This study will include 10 female breast cancer survivors and 10 male prostate cancer survivors. For the first 12 weeks on study (Part 1), participants will train with an exercise physiologist (EP) for 150 minutes/week. This training will be delivered by web-based video conferencing. For the next 12 weeks (Part 2), participants will be instructed to do patient-directed exercise.

ELIGIBILITY:
Inclusion Criteria:

* Male previously diagnosed with prostate cancer or female previously diagnosed with breast cancer.
* For breast cancer, minimum of 3 months post-active treatment completion. Active treatment includes chemotherapy, biologic therapy, radiation therapy, surgery, and any combination. Long-term hormonal/biologic treatments are acceptable.
* For prostate cancer, minimum of 3 months post-active treatment completion. Active treatment includes chemotherapy, biologic therapy, radiation therapy, surgery, and any combination. Long-term hormonal/biologic treatments are acceptable, except for androgen receptor-targeted therapies (such as enzalutamide, apalutamide, darolutamide, or abiraterone). Patients currently on active surveillance are eligible even if they have not received prior anti-cancer treatment.
* Has access to tablet, laptop, or desktop computer with video capabilities connected to the internet with a screen at least 13 inches across.
* Physically able to complete modified Bruce submaximal treadmill test, leg strength test, grip strength test, and InBody per patient self-assessment.
* Physician clearance to participate in this study. Can be done through review of patients' medical records.
* Ability to read, write, and understand English.
* Has a chair at home to use for exercise that is not on wheels and has a solid back (not a reclining chair).
* Ambulatory without assistance.
* Has a clear 5 x 6-foot space at home in which to exercise.
* Age >18 years.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Active treatment planned within the next 6 months. Active treatment includes chemotherapy, biologic therapy, radiation therapy, surgery, and any combination. Long-term hormonal/biologic treatments are acceptable, except for AR-targeted therapies for prostate cancer.
* Known metastatic disease.
* Grade 3 or higher peripheral neuropathy.
* Major surgery within 3 months of baseline visit.
* Positive pregnancy test for women of child-bearing potential.
* Answers yes to any question on the Physical Activity Readiness Questionnaire unless study participation is cleared by a physician.
* Known allergy to Fitbit device.
* Currently meeting physical activity guidelines (score of >23 on Godin-Shephard Leisure-Time Physical Activity Questionnaire).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Attendance | 12 weeks
  Explore adherence to intervention delivery measured through attendance (frequency of Skype sessions attended and fully completed)
Adherence | 12 weeks
  Explore adherence to intervention delivery measured through retention (participation from baseline through final assessment)
Patient consent | 1 day
  Explore adherence to intervention delivery measured through percentage of patients approached who sign consent
Manipulation check | 12 weeks
  Explore adherence to intervention delivery measured through scores on manipulation check after each session (2 questions asked by exercise physiologist on sound and visual clarity of the session)

SECONDARY OUTCOMES:
Changes in oxygen uptake (baseline - mid-study visit) | 12 weeks
  Change in vO2 submax measurement (rate of oxygen uptake during exercise) between baseline & mid-study visits as measured by Bruce submaximal treadmill test.
Changes in oxygen uptake (mid-study visit - end of study visit) | 12 weeks
  Change in vO2 submax measurement (rate of oxygen uptake during exercise) between mid-study & end of study visits as measured by Bruce submaximal treadmill test.
Changes in oxygen uptake (baseline - end of study visit) | 24 weeks
  Change in vO2 submax measurement (rate of oxygen uptake during exercise) between baseline & end of study visits as measured by Bruce submaximal treadmill test.
Changes in strength test (baseline - mid-study visit) | 12 weeks
  Change in muscle strength measurement between baseline & mid-study visits as measured by grip strength test and leg press.
Changes in strength test (mid-study visit - end of study visit) | 12 weeks
  Change in muscle strength measurement between mid-study & end of study visits as measured by grip strength test and leg press.
Changes in strength test (baseline - end of study visit) | 24 weeks
  Change in muscle strength measurement between baseline & end of study visits as measured by grip strength test and leg press.
Changes in resting heart rate (baseline - mid-study visit) | 12 weeks
  Changes in resting heart rate between Baseline & mid-study visits
Changes in resting heart rate (mid-study visit - end of study visit) | 12 weeks
  Changes in resting heart rate between mid-study & end of study visits
Changes in resting heart rate (baseline - end of study visit) | 24 weeks
  Changes in resting heart rate between Baseline & end of study visits
Changes in body composition (baseline - mid-study visit) | 12 weeks
  Changes in body composition between baseline & mid-study visits as measured by InBody (non-invasive body composition analysis that calculates weight, skeletal muscle mass, fat mass, BMI, and body fat percent using Bio-Electrical Impedance Analysis).
Changes in body composition (mid-study visit - end of study visit) | 12 weeks
  Changes in body composition between mid-study & end of study visits as measured by InBody (non-invasive body composition analysis that calculates weight, skeletal muscle mass, fat mass, BMI, and body fat percent using Bio-Electrical Impedance Analysis).
Changes in body composition (baseline - end of study visit) | 24 weeks
  Change in body composition between baseline & end of study visits as measured by InBody (non-invasive body composition analysis that calculates weight, skeletal muscle mass, fat mass, BMI, and body fat percent using Bio-Electrical Impedance Analysis).
Subjective impact | 24 weeks
  Subjective impact of exercise intervention as measured by changes in participant-reported rating of exercise self-efficacy and intentions to remain active

CONTACTS AND LOCATIONS:
Overall Officials: Celina Shirazipour, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States